CLINICAL TRIAL: NCT01646645
Title: A Phase II Trial of Primary Transplant Donor Derived CMVpp65 Specific T-cells for The Treatment of CMV Infection or Persistent CMV Viremia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Primary Transplant Donor Derived CMVpp65 Specific T-cells for The Treatment of CMV Infection or Persistent CMV Viremia After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-086
Expanded Access: NCT03010332 (No longer available)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-10

CONDITIONS: Cytomegalovirus
Keywords: CMVpp65 specific T-cells; Stem Cell Transplantation; 12-086

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group I (Experimental): This is a single-arm non-randomized single institution phase 2 trial, designed to evaluate the therapeutic activity of CMVpp65-CTLs generated from seropositive HSCT donors when adoptively transferred into transplant recipients with persistent CMV infection or viremia. Patients eligible for this trial will be consenting recipients of related or unrelated HSCT who have an active CMV infection or persistent CMV viremia for ≥ 2 weeks despite treatment with anti-viral agents or who cannot be maintained on anti-viral therapy due to treatment related toxicity.
  Interventions: Biological: CMV-pp65 CTLs

INTERVENTIONS:
Biological: CMV-pp65 CTLs — Patients will be treated with CMVpp65-CTLs derived from their transplant donor. These will be patients with CMV seropositive transplant donors who have previously provided leukocytes for generation of CMVpp65-CTL and for whom such CMVpp65-CTL are available. The T-cells to be infused will be selected based on criteria mentioned in section 4.0 from our bank of GMP grade CMVpp65-CTL. T-cells will be administered by bolus intravenous infusion. In this phase II trial, patients will be treated at doses of 1 x 106 CMVpp65-CTL/kg/dose/week for 3 weeks. Patients will be observed for the following 3 weeks. Additional 3 week courses of CMVpp65-CTL may be administered if levels of CMV DNA in blood are still detectable despite disease stabilization or improvement.

SUMMARY:
The purpose of this study is to see how well transfusions of T-cells work in treating CMV. T-cells are a type of white blood cell that helps protect the body from infection. A transfusion is the process by which blood from one person is transferred to the blood of another. In this case, the T-cells are made from the blood of donors who are immune to CMV. The T-cells are then grown and taught to attack the CMV virus in a lab.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must satisfy at least one of the following criteria:

  1. The patient must have a clinically documented condition associated with CMV (e.g. interstitial pneumonia, hepatitis, retinitis, colitis) Or
  2. The patient must have microbiological evidence of CMV viremia or tissue invasion as attested by viral culture, or detection of levels of CMV DNA in the blood or body fluids consistent with CMV infection.

Patient must also satisfy at least one of the following criteria:

1. The patient's CMV infection is clinically progressing or CMV viremia is persistent or increasing (as evidenced by quantitation of CMV DNA in the blood) despite two weeks induction therapy with antiviral drugs.

   Or
2. The patient has developed CMV viremia as attested by viral culture, or detection of levels of CMV DNA in blood or body fluids while receiving prophylactic doses of antiviral drugs to prevent CMV infection post transplant.

Or c. The patient is unable to sustain treatment with antiviral drugs due to drug associated toxicities (e.g. myelosuppression [ANC< 1000μl/ml without GCSF support] or nephrotoxicity [corrected creatinine clearance ≤ 60 ml/min/1.73 m2 or serum creatinine > 2 mg/dl]) Patient has CMV specific T-cells from the donor of his/her HSCT available. CMV infections are life threatening, and may involve multiple organ systems such as the lungs, liver, gastrointestinal tract, hematopoietic and central nervous systems. Antiviral drugs used for treatment may also compromise renal and hematopoietic function. Therefore, dysfunctions of these organs will not affect eligibility for this protocol Patients must meet the following clinical criteria to receive CMVpp65-CTL infusions

1. Stable blood pressure and circulation, not requiring pressor support
2. Evidence of adequate cardiac function as demonstrated by EKG and/or echocardiography.
3. A life expectancy of at least 3 weeks, even if requiring artificial ventilation.
4. There are no age restrictions

Exclusion Criteria:

* Patients requiring high doses of glucocorticosteroids (≥ 0.3 mg/kg prednisone or its equivalent) 2. Patients who are moribund 3. Patients with other conditions not related to CMV infection (e.g. uncontrolled bacterial sepsis or invasive fungal infection) which are also life-threatening and which would preclude evaluation of the effects of a T-cell infusion.

3.4. Patients who are pregnant 6.1.3 Donor Inclusion Criteria 6.1.3a Donors in Group 1 (Historical Donors) Donors in Group 1 (Section 5.1) would have already been determined to be eligible and will have donated blood or leukocytes to establish CMV-specific T-cells under IRB # 05-065, 07-055, 95-024, or 11-130. There are no additional eligibility requirements for these donors.

6.1.3b Donors in Groups 2 & 3 (Prospective and Volunteer Donors)

Transplant donors and healthy HLA typed volunteers who agree to provide T-cells for Third-party donation (section 5.1, Groups 2 and 3) will need to meet the following eligibility requirements prior to donation:

1. Donors must satisfy the criteria specified in FDA 21 CFR 1271.
2. Donors must be typed for HLA-A, B, C and DR
3. Donors must have a hemoglobin value > 10g/dl
4. Donors must be capable of undergoing, at least, a single standard 2 blood volume leukapheresis or a donation of one unit of whole blood

6.1.4 Donor Exclusion Criteria

1. HTLV/HIV(+) or Hepatitis B or C antigen(+) donors
2. Donors who are known CMV seronegative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Prockop, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I
Started | 58
Completed | 28
Not Completed | 30
Not completed — No Treated | 1
Not completed — Inevaluable Donor | 29

BASELINE CHARACTERISTICS:
Arm/Group | Group I
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 49 [1 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response
Description: The endpoint of this study is complete response, defined as the clearance of the CMV infection 3-7 weeks following completion of the last cycle of CMV CTLs. The evaluation of treatment efficacy will be assessed separately for patients receiving CMV specific T cells from their transplant donor.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I
Number analyzed (Participants) | 58
Participants
  Participants With Complete Response | 8
  Participants Without Complete Response | 50

2. Primary Outcome: Number of Participants With Toxicities
Description: For the evaluation of toxicities, the NCI Standard Toxicity Scale 4.0 will be employed.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Group I
Number analyzed (Participants) | 58
participants | 58

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Group I
All-Cause Mortality (participants affected / at risk) | 18/58
Serious Adverse Events (participants affected / at risk) | 11/58
Other Adverse Events (participants affected / at risk) | 28/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=58)
Acidosis (Metabolism and nutrition disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Catheter related infection (Infections and infestations) | 2
Death NOS (General disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Neutrophil count decreased (Investigations) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=58)
Platelet count decreased (Investigations) | 20
Lymphocyte count decreased (Investigations) | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 13
Neutrophil count decreased (Investigations) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 12
White blood cell decreased (Investigations) | 10
Hypermagnesemia (Metabolism and nutrition disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 4
Alkaline phosphatase increased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT01646645/Prot_SAP_000.pdf